CLINICAL TRIAL: NCT00157612
Title: A Randomized Control Trial of a Clinical Pathway for Nursing Home Pneumonia.
Brief Title: A Clinical Pathway for Nursing Home Acquired Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00-1848; long term care (Other: McMaster University)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Pneumonia; Lower Respiratory Tract Infection
Keywords: pneumonia; lower respiratory tract infection; clinical pathway; nursing home; long-term care; randomized control trial
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Other): use of oral anti-microbials, portable chest radiographs, oxygen saturation monitoring, re-hydration and close monitoring by a research nurse
  Interventions: Procedure: a clinical pathway nursing home acquired pneumonia
- Comparator (No Intervention): usual care

INTERVENTIONS:
Procedure: a clinical pathway nursing home acquired pneumonia — treatment in nursing homes according to a clinical pathway, which included use of oral anti-microbials, portable chest radiographs, oxygen saturation monitoring, rehydrations and close monitoring by research nurse
  Other Names: Nursing Home Residents with Pneumonia
  Arms: Intervention

SUMMARY:
Nursing home residents are frequently transferred to hospital for management of pneumonia. This often leads to hospital related complications and is a burden on the acute care health system. The purpose of this study is to assess whether managing residents with pneumonia and lower respiratory tract infection on site in the nursing home can reduce hospital admissions and can reduce complications and improve quality of life for residents. We have randomized residents with nursing home acquired pneumonia to on-site management, using a clinical pathway, versus usual care.

DETAILED DESCRIPTION:
We conducted a cluster-randomized controlled trial where nursing homes were randomized to either use of a clinical pathway or usual care for management of nursing home acquired pneumonia. The clinical pathway included chest radiographs performed on-site in the nursing home by a mobile x-ray unit, use of hypodermocylysis (subcutaneous infusion) for re-hydration, administration of an oral antimicrobials, and use of pulse oximetry to assess oxygenation. The main outcomes were hospital admission rate and length of stay. Secondary outcomes included health related quality of life, rates of both infectious and non-infectious complications within four weeks of onset of symptoms; mortality rate of residents with pneumonia (death from all causes within 30 days of onset of symptoms. Time to stabilization of vital signs, as well as functional status at four weeks, were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms or signs of lower respiratory tract infection as defined by standardized criteria.

Exclusion Criteria:

* Residents were excluded if they were not expected to live longer than 30 days from the date of enrollment, had a previous anaphylactic or serious allergic reaction to quinolones, had advanced directives that they are not be transferred to hospital for treatment.

Min Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2001-01; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Hospital admission, length of stay

SECONDARY OUTCOMES:
Health related quality of life,
complication rates,
mortality,
functional status,
time to stabilization of vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Loeb, MD MSc FRCPC, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Loeb M, Carusone SC, Goeree R, Walter SD, Brazil K, Krueger P, Simor A, Moss L, Marrie T. Effect of a clinical pathway to reduce hospitalizations in nursing home residents with pneumonia: a randomized controlled trial. JAMA. 2006 Jun 7;295(21):2503-10. doi: 10.1001/jama.295.21.2503. PMID 16757722